CLINICAL TRIAL: NCT05406869
Title: A Prospective, Multicenter, Single-arm Study to Evaluate the Safety and Efficacy of Pulsed Sonic Balloon Dilatation Catheter and Pulsed Sonic Generater in the Treatment of Coronary Calcified Lesions
Brief Title: Clinical Trials of Pulsed Sonic Balloon Dilatation Catheter and Pulsed Sonic Generater
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP-Pulsed Sonic Balloon-2022
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Coronary Calcified Disease
Keywords: Coronary Sonic Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulsed sonic balloon dilatation catheter and pulsed sonic generater (Experimental): All subjects will receive treatment from the pulsed sonic balloon dilatation catheter
  Interventions: Device: Pulsed Sonic Balloon Dilatation Catheter and Pulsed Sonic Generater

INTERVENTIONS:
Device: Pulsed Sonic Balloon Dilatation Catheter and Pulsed Sonic Generater — Deliver Pulsed Sonic Balloon Dilatation Catheter to the target vessel prior to placing a coronary stent or others

SUMMARY:
The prospective, multicenter, single- arm study is designed to verify the safety and efficacy of pulsed sonic balloon dilatation catheter and pulsed sonic generater in the treatment of coronary calcification lesions.

DETAILED DESCRIPTION:
The study will include a total of 170 patients with calcified coronary lesions who will be treated with pulsed sonic balloon dilatation catheter and pulsed sonic generater. Optical coherence tomography (OCT) imaging subgroups of 30 patients were designed in 1-2 centers to further accurately assess the treatment effect of calcified lesions.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤age≤80 years old, males or females;
2. Life expectancy ≥ 6 months;
3. Patients with evidence of asymptomatic myocardial ischemia, stability or instability; with angina, or obsolete heart infarction for interventional therapy;
4. The target lesion is primary, in situ coronary artery lesion;
5. The target vessel reference diameter is 1.5-4.0mm, and the lesion length is ≤40mm (visual inspection);
6. Target lesion is with a visually estimated stenosis of ≥70%(or≥50% with evidence of myocardial ischemia) ;
7. Highly calcified lesions;
8. Only one target lesion requiring sonic balloon treatment is allowed;
9. The number of non-target lesions requiring interventional treatment is no more than 2, and the target lesions should be treated after the non-target lesions are successfully treated;
10. Patients who can understand the purpose of the trial, voluntarily participate and sign the informed consent form, and can accept required clinical follow-up.

Exclusion Criteria:

1. New York Heart Association (NYHA) class III or IV;
2. Severe liver and kidney damage, transaminase more than 3 times the upper limit of normal, creatinine > 2.5mg/dL (221μmol/L) or chronic renal failure requiring long-term dialysis;
3. Stroke occurred within 6 months of joining the group, excluding transient is chemic attack (TIA) and cavity infarction;
4. Have a history of active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months of joining the group;
5. Platelet count <80×10⁹/L;
6. Subject refuses or is not suitable for CABG surgery;
7. The target lesion is planned to undergo coronary atherectomy, laser, double guide wire balloon, mastoid balloon, cutting balloon or thrombus aspiration;
8. Dissection of the target vessel after preoperative angiography or guide wire pass through;
9. The stent has been implanted within 10mm of the proximal or distal end of the target lesion, and there is a definite or possible thrombus in the target vessel;
10. The target lesion is located or involved within 5mm of the opening of LAD, LCX and RCA;
11. Left main stem disease or bridge vascular disease;
12. Angiography shows that the blood vessel path is tortuous, and the test device is difficult to reach the target position or difficult to recover;
13. Patients with implanted pacemakers or cardiac rhythm devices;
14. Evidence of aneurysm within 10 mm of the target lesion;
15. Patients who are known to be allergic to heparin, contrast agents, aspirin, clopidogrel, and anesthetics;
16. The subject is currently participating in another drug or device clinical study that has not yet completed;
17. Pregnant or nursing subjects;
18. Other patients should be excluded based on the assessment of the investigators;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-10-07 (Estimated); Study Completion 2023-01-07 (Estimated)

PRIMARY OUTCOMES:
Procedural success rate | immediate post-procedure
  Procedural success was defined as residual stenosis ≤30% after successful stent delivery without the occurrence of in-hospital adverse cardiac events (include cardiac death, target vessel-related myocardial infarction (TV-MI) and target lesion revascularizition)

SECONDARY OUTCOMES:
Device success rate | immediate post-procedure
  Device success was defined as residual stenosis ≤50% with the successful delivery, deployment and withdrawal of pulsed acoustic wave balloon dilatation catheter to the target lesion.
Lumen diameter obtained | immediate post sonic balloon treatment, immediate post-procedure
  Defined as the change of minimal luminal diameter[MLD] between the Follow-up points and baseline.
Percentage of diameter stenosis | immediate post sonic balloon treatment, immediate post-procedure
  Defined as (1-minimal luminal diameter[MLD]/reference vessel diameter[RVD])*100%
Target Lesion Failure (TLF) | before discharge or 7 days post-procedure, 30 days post-procedure
  Target lesion failure is a composite endpoint of cardiac death, target vessel related myocardial infarction (TV-MI) and the ischemia-driven target lesion revascularization.
Patient-related cardiovascular clinical composite endpoint (POCE) | before discharge or 7 days post-procedure, 30 days post-procedure
  Including all-cause death, all MI, or any revascularization
Confirmed and probable thrombotic events | before discharge or 7 days post-procedure, 30 days post-procedure
  Including Acute thrombosis, Early thrombosis, Late thrombosis, Very late thrombosis.
The stability of the pulse sonic energy generator | immediate post-procedure
  Including excellent, good and poor levels
Ease of use of pulsed acoustic energy generators | immediate post-procedure
  Including excellent, good and poor levels

CONTACTS AND LOCATIONS:
Overall Officials: Yida Tang, Study Chair — Peking University Third Hospital
Locations (14):
- China (14):
  - Beijing Anzhen Hospital, Capital Medical Univesity, Beijing, Beijing Municipality
  - Beijing Chao-yang Hospital , Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Southwest Hospital of Amu, Chongqing
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The Second Xiangya Hospital of Central South University, Hunan
  - Xiangya Hospital Central South University, Hunan
  - LinFen Central Hospital, Shanxi
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Xuzhou central hospital, Xuzhou
  - Sir Run Run Shaw Hospital ZheJiang University School of Medicine, Zhejiang